CLINICAL TRIAL: NCT05068089
Title: Health, Economic Analysis and Clinical Aspects of a Pediatric Cohort With Severe Motor and Intellectual Disabilities in Enteral Nutrition With Dedicated Formula. A Case-control Retrospective Observational Study for the Management of Gastroesophageal Reflux: the Role of Fundoplication According to Nissen.
Brief Title: Health, Economic Analysis and Clinical Aspects of Patients With Neurological Disabilities in Enteral Nutrition With Dedicated Formula. The Role of Nissen's Fundoplication in the Management of Gastroesophageal Reflux
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: Nestlé Health Science Spain (Industry)
Responsible Party: Sponsor
Other Study IDs: 2322_Opbg_2021
Record Dates: First submitted 2021-09-14; First posted 2021-10-05 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Gastro-Esophageal Reflux; Fundoplication
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication; Enteral Nutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nissen fundoplication surgery and Enteral nutrition: The cohort population retrospectively enrolled in the study is represented by pediatric patients with severe motor and intellectual disabilities (with progressive e non- progressive neurological disease) followed-up at Nutrition Unit of Ospedale Pediatrico Bambino Gesù between January 2009 to January 2020.
  Interventions: Procedure: Nissen fundoplication; Biological: Enteral nutrition

INTERVENTIONS:
Procedure: Nissen fundoplication — Nissen fundoplication, numbers, reasons and length of hospitalizations, gastrointestinal symptoms and survival
Biological: Enteral nutrition — Type and switch of enteral nutrition formula (tube, PEG, PEJ)

SUMMARY:
Nutritional difficulties are common in children with neurodisabilities and can be associated with malnutrition and gastrointestinal diseases, such as gastro-esophageal reflux disease (GERD) and constipation. Neurological disorders can be divided into two main categories: progressive (neurodegenerative, mitochondrial disease) and non-progressive (cerebral palsy) neurodisabilities; nature of the disorders can impair on the nutritional status of these children. In 2017, ESGHAN published guidelines with specific nutritional claims. Approximately 46%-90% of children with neurodisabilities suffer from malnutrition and an enteral feeding is necessary to reach the nutritional requirements. In addition, a relevant issue for these children is GERD, reaching up to 70% prevalence. The treatment of GERD could be based on pharmacological therapy (protonic pomp inhibitor, PPI), on nutritional treatment (changing type of formula) or on surgical treatment (Nissen Fundoplication). European guidelines for GERD recommend PPI as the first line, with fundoplication being considered in cases of failure of optimized medical therapy. Enteral feeding can be considered in order to avoid malnutrition and is justified when other efforts to increase nutritional intake. Enteral feeding can be provided by nasal tube at the beginning, but a gastrostomy feeding tube would be preferred for a long-term nutrition (greater than six weeks). A jejunal tube can be introduced through the gastrostomy; jejunal feeding is appropriate in patients with recurrent vomiting and/or tube feeding-related aspiration, severe gastroesophageal reflux, and gastroparesis. Different types of formulas can be used for enteral nutrition and can be offered by nasal tube, percutaneous endoscopic gastrostomy (PEG) or percutaneous endoscopic jejunostomy (PEJ). Whey-based formulas have been shown to empty from the stomach more rapidly than casein-based formulas, which may be helpful for patients presenting with delayed gastric emptying. Use of peptide-based, 100% whey protein formulas are associated with improved feeding tolerance, increased consistency in meeting nutritional needs, and a reduction in gastrointestinal issues associated with vomiting and aspiration of feeds. For these reasons, the aim of this study is to retrospectively evaluate the role of different formulas against Nissen fundoplication, regarding tolerance, utility, applicability and safeness of these products, by performing a cost analysis.

DETAILED DESCRIPTION:
Nutritional difficulties are common in children with severe motor and intellectual disabilities (SMID) and can be associated with malnutrition, growth difficulties, micronutrient deficiencies, osteopenia and nutritional comorbidities. In children with SMID, neurological disorders can be divided into two main categories: progressive and non-progressive neurodisabilities. Progressive neurological disorders feature a progressive decline of functioning, which can occur over many years and decades, or more rapidly over weeks and months. Such disorders include mitochondrial disorders, myopathies, disorders only involving the spinal cord, or neuromuscular disorders and are likely to have a lifelong course. On the other hand, non-progressive neurological disorders apparently do not feature a progression of disease, as seen in the most common condition, infantile cerebral palsy (ICP).

Both progressive and non-progressive neurological disorders feature nutritional difficulties following involvement of the central nervous system or neuromuscular disorders. In patients with both conditions, oral motor dysfunction (involving tongue, chin or the whole mouth) results in the development of feeding problems.

Moreover, gastrointestinal disturbances in these children reflect the interplay between the central nervous system and the enteric nervous system.

In 2017, specific guidelines for the nutritional management of children with neurological disease were published by the ESPGHAN. These guidelines mention the following five warning signs ("red flags") for the identification of nutritional issues in children with neurological impairment: (1) physical signs of undernutrition (decubitus skin problems, poor peripheral circulation), (2) weight for age Z-score <-2, (3) triceps skinfold thickness <10th centile forage and sex, (4) mid-upper arm fat or muscle area <10thcentile and (5) faltering weight and/or failure to thrive.

Guidelines also suggest not to limit nutritional status assessment based on weight and height alone, but to also perform evaluation of knee height or tibial length when height cannot be measured, of fat mass by skinfold thickness, of BMD by DXA scans, and of micronutrient status.

Malnutrition is a relevant issue for children with SMID, with a reported 46%-90% prevalence and multifactorial etiology, including inadequate dietary intake; gastro-oesophageal reflux disease (GERD); constipation; underlying neurological disability and relevant medications, including antiepileptic drugs. More in detail, GERD in children with SMID is a well-described phenomenon, reaching up to 70% prevalence and potentially resulting in aspiration pneumonia and fatal outcomes. In these patients, GERD occurs as a result of impaired motility of esophagus and the lower esophageal sphincter (LOS), which lead to the development of retrograde, regurgitation of gastric contents into the esophagus.

On top of the underlying neurological impairment causing delayed gastric emptying and altered esophageal motility, several other factors are involved, such as increased abdominal pressure secondary to scoliosis, constipation and spasticity of abdominal musculature. As also suggested by ESPGHAN, several diagnostic procedures should be considered to objectively investigate GERD in children with neurological impairments (NI), such as upper GI endoscopy and/or esophageal pH- or pH/multichannel intraluminal impedance monitoring. As GERD is highly prevalent, it can be useful to consider a short trial with PPIs: these drugs should be considered as the first-line treatment, while use of prokinetic agents should be limited owing to the weaker efficacy and higher incidence of side effects.

Several treatments are available for GERD, including enteral mixtures containing whey proteins; surgical treatments (Fundoplication according to Nissen, NF) are also available.

Enteral nutrition should be considered only following failure of other strategies aimed to increase nutritional intake in order to reduce the risk of malnutrition. Children with NI should preferably be provided long-term nutritional support by a gastrostomy feeding tube, with gastrostomy to be reserved for cases in which enteral feeding is supposed to last more than six weeks), or to increase weight, improve overall health and decrease feeding times for children with neurological impairment. Caregivers might similarly have a beneficial effect for quality of life. Laparotomy, laparoscopy or endoscopy can all be used for the placement of a gastrostomy tube, with percutaneous endoscopic gastrostomy (PEG) being at present the most favored procedure. Tube placement, however, carries several risks, including infection, perforation, bleeding, tube migration/dislocation, intestinal fistulas and obstruction. Over time, the presence of a gastrostomy tube might lead to the development, or to the progression to more severe forms of GERD.

Another viable choice for patients who already have a gastrostomy is the placement of a jejunal tube through the gastrostomy itself. However, as these tubes can migrate back to the stomach or can incur tube obstruction or mechanical failure, jejunal tubes require careful monitoring. Additionally, use of a jejunal tube should be considered only for patients who cannot use other forms of enteral feeding, such as recurrent vomiting and/or tube feeding-related aspiration, severe gastroesophageal reflux, and gastroparesis. Favorable clinical outcomes were found following the use of combined gastric decompression via PEG and simultaneous jejunal nutrition.

Independently of the strategy used (tube feeding, PEG or PEJ), several formulations are available, most for which provide 1-2 kcal/ml, with or without fibre.

ESPGHAN recommendations state that standard (1.0 kcal/mL) polymeric age-appropriate formula including fiber should be used for children with NI older than 1 year, a high energy density formula (1.5 kcal/mL) containing fiber in cases of poor volume tolerance and human milk, a standard infant formula, or nutrient dense infant enteral formula as clinically indicated in infants. Moreover, a low-fat, low-calorie, high-fiber, and micronutrient replete formula for the maintenance of enteral tube feeding after nutritional rehabilitation in immobile children is recommended; and using a trial of whey-based formula in cases of gastroesophageal reflux, gagging, and retching in children with NI.

Patients with delayed gastric emptying can have beneficial effects from whey-based formulas, which based on the more rapid emptying than casein-based formulas. Additionally, some populations might be preferentially treated with hydrolyzed over intact proteins. Feeding tolerance is improved by the use of peptide-based, 100% whey protein formulas, and similarly other beneficial effects, such as increased compliance to meeting nutritional needs and reduction of gastrointestinal complications secondary to vomiting and feed aspiration, have been reported. Patients with gastrointestinal illnesses, including pancreatic insufficiency or malabsorption, should preferentially be treated with peptide-based diets, which can also be useful for children with developmental delays in the absence of a definite diagnosis of gastrointestinal impairment.

Medical management of GERD in NI children has historically been burdened by low compliance, leading to the widespread use of surgical treatments such as a Nissens, Thal, Toupet or Belsey fundoplication to provide relief from reflux. The fundoplication procedure is performed by wrapping the stomach fundus around the gastro-oesophageal junction, therefore creating an additional barrier to acid reflux: more in detail, the procedures involves correction of hiatal herniation, lengthening of the intra-abdominal portion of the oesophagus, and tightening of the crura, therefore increasing pressure at the LOS level. According to the different extent of the operation, fundoplication procedures can provide both a full 360° wrap and a partial 180° wrap. Fundoplication, however, has other consequences, such as increasing the risk of vagal nerve damage which in turn can elicit the emetic reflex, or promoting the onset of seizures or pulmonary disease secondary to increased abdominal pressure or to the surgery itself. Other surgery-related complications include gas bloat syndrome, impaired gastric accommodation, gastric hypersensitivity, rapid gastric emptying (or 'dumping syndrome'), retching or dysphagia. Additionally, as NI children often have other underlying conditions, such as epilepsy or scoliosis, the risk of failure of any anti-reflux intervention should be considered: in these children, fundoplication has a high failure rate, reaching up to 40%, and significant morbidity and mortality, with a 1% to 3% mortality rate. Reflux might persist following fundoplication in about 12% to 30% of children with NI, and almost two-thirds of treated children (59%) develop postoperative complications.

It is therefore unsurprising that ESPGHAN recommendations state that fundoplication should be only considered in children with NI following failure of optimized medical therapy for GERD. Indeed, beneficial effects can be obtained by anti-reflux surgery in children with confirmed GERD who did not have clinical improvement despite adequate medical treatment, or who require long treatment duration, who are non-compliant to medical therapy, or who have life-threatening complications of GERD. Following failure of medical treatment, surgery is most likely beneficial in children with asthma, recurrent aspiration, or other GERD-related respiratory complications. If medical treatment achieves its target of controlling symptoms, there is supposedly no additional benefit from antireflux surgery, also owing to the aforementioned risks.

The choice of treatment is based on clinical considerations which may vary between patient and patients. The ESPGHAN guidelines recommend making a careful diagnosis of possible causes and prescribing nutritional adaptation and therapeutic treatments (proton pump inhibitors, PPIs) as first-line approaches, considering Nissen surgery only in case of failure of medical therapy / nutritional.

In conclusion, the clinical management of children with neurological impairments could be variable.

As shown, enteral nutrition through specific formulas seems to be well tolerated and seems to reduce gastro-intestinal (GI) intolerance in children with impaired neurological functions. From literature it can be said that from a clinical point of view, enteral nutrition based on whey proteins can be considered a valid alternative to NF, reducing not only the incidence of GI intolerance symptoms but also the need for further health interventions.

Despite these findings, no data are available in literature regarding a comparison between special formula and Nissen fundoplication and the main aims of this study is to fill this evidence's gap.

Based on evidences showing that a changing from an intact protein enteral feeding to a 100% whey, peptide-based formula improved the feeding tolerance, the hypothesis that peptide-based formula could be comparted to NF turns out to be the next step in the analysis of these products. In this way, it might be useful to evaluate the role of different formulas against NF, regarding tolerance, utility, applicability and safeness of these products.

This study was been designed as a monocentric, retrospective observational (cohort) study with the aim to carry out a healthcare cost analysis between patients undergoing NF surgery and patients treated with whey protein-based enteral nutrition.

By performing this cost analysis, it may be possible to evaluate the better timing for Nissen Fundoplication surgery in patient with enteral nutrition and secondary, it may be possible to describe and to quantify resource consumption and the occurrence of GI disorders related to the different types of formulas.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe motor and intellectual disabilities (SMID);
* Pediatric patients ( 29 days; <18 years);
* Subjects whose enteral nutrition through a nasogastric tube or endoscopic gastrostomy; percutaneous (PEG) involves the administration of a special formula based on whey protein or a formula based on caseinates;
* Subjects undergoing or not NF surgery.

Exclusion Criteria:

* Patients less than 24 months of follow-up at the closing of the database;
* Patients with less than 12 months of observation.

Ages: 29 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes children with neurological damage (0-18 years) treated in the Nutritional Clinic Department from January 2009 to January 2020 due to nutritional problems and food and / or gastrointestinal intolerances.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
To identify the annual economic impact related to the treatment of patients undergoing NF surgery and the costs related to patients undergoing enteral nutrition, analyzing type of formula offered. | 11 years
  Annual economic impact expressed in Euro, calculated by Health Direction based on specific invoice (SDO) and specific calculator (provided by Italy Ministry of Health); length of hospitalization expressed in days

SECONDARY OUTCOMES:
To evaluate whether the need for NF is postponed or reduced in the patient population fed with enteral formulas based on whey proteins | 11 years
  Time (expressed in days) between the onset of enteral nutrition and the need to carry out the surgery for NF
Describe and quantify the occurrence of GI disorders associated with different types of enteral nutritional formulas (whey protein vs caseinates) | 11 years
  Number of participants with new onset of GI disorders according to treatment group (whey protein vs caseinates); number of patients with persistent GI disorders according to treatment group (whey protein vs caseinates). ; Number of participants with remitting GI disorders according to treatment group (whey protein vs caseinates).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS, Ospedale Pediatrico Bambino Gesù, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
Only the publication article will be shared with other researchers.

REFERENCES:
- [Background] Romano C, van Wynckel M, Hulst J, Broekaert I, Bronsky J, Dall'Oglio L, Mis NF, Hojsak I, Orel R, Papadopoulou A, Schaeppi M, Thapar N, Wilschanski M, Sullivan P, Gottrand F. European Society for Paediatric Gastroenterology, Hepatology and Nutrition Guidelines for the Evaluation and Treatment of Gastrointestinal and Nutritional Complications in Children With Neurological Impairment. J Pediatr Gastroenterol Nutr. 2017 Aug;65(2):242-264. doi: 10.1097/MPG.0000000000001646. PMID 28737572
- [Background] Hasegawa M, Tomiwa K, Higashiyama Y, Kawaguchi C, Kin H, Kubota M, Shima M, Nogami K. Risk factors of malnutrition in children with severe motor and intellectual disabilities. Brain Dev. 2020 Nov;42(10):738-746. doi: 10.1016/j.braindev.2020.06.009. Epub 2020 Jul 2. PMID 32624241
- [Background] van den Engel-Hoek L, de Groot IJ, de Swart BJ, Erasmus CE. Feeding and Swallowing Disorders in Pediatric Neuromuscular Diseases: An Overview. J Neuromuscul Dis. 2015 Nov 20;2(4):357-369. doi: 10.3233/JND-150122. PMID 27858755
- [Background] Sullivan PB. Gastrointestinal disorders in children with neurodevelopmental disabilities. Dev Disabil Res Rev. 2008;14(2):128-36. doi: 10.1002/ddrr.18. PMID 18646021
- [Background] Savage K, Kritas S, Schwarzer A, Davidson G, Omari T. Whey- vs casein-based enteral formula and gastrointestinal function in children with cerebral palsy. JPEN J Parenter Enteral Nutr. 2012 Jan;36(1 Suppl):118S-23S. doi: 10.1177/0148607111428139. PMID 22237871
- [Background] Minor G, Ochoa JB, Storm H, Periman S. Formula Switch Leads to Enteral Feeding Tolerance Improvements in Children With Developmental Delays. Glob Pediatr Health. 2016 Dec 21;3:2333794X16681887. doi: 10.1177/2333794X16681887. eCollection 2016. PMID 28229094